CLINICAL TRIAL: NCT02417220
Title: Weight Watchers Online 2015
Acronym: WWO 2015
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: WW International Inc (Industry); University of Tennessee (Other)
Responsible Party: Principal Investigator, John Graham Thomas, Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WeightWatchersOnline2015
Record Dates: First submitted 2015-04-08; First posted 2015-04-15 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Obesity; Overweight; Body Weight
MeSH Terms: conditions — Obesity; Overweight; Body Weight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight Watchers Online 2015 (Active Comparator)
  Interventions: Behavioral: Weight Watchers Online 2015 Program
- Weight Watchers Online 2015 Enhanced (Experimental)
  Interventions: Behavioral: Weight Watchers Online 2015 Program; Other: Electronic Scale with Feedback

INTERVENTIONS:
Behavioral: Weight Watchers Online 2015 Program — Access to the Weight Watchers Online 2015 program available via the Internet on personal computers, tablet computers, and/or smartphones already owned by participants.
Other: Electronic Scale with Feedback — Provision of an electronic scale that automatically transmits body weights to the Weight Watchers Online 2015 program, which generates a weekly feedback message on weight loss progress.
  Arms: Weight Watchers Online 2015 Enhanced

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial to compare the weight losses produced by the Weight Watchers Online program revised for 2015 (WWO2015) and WWO2015 plus the provision of an electronic scale and weekly email feedback on weight loss (WWO2015 Enhanced), over a 6-month period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Body mass index (BMI) between 27 and 40 kg/m2
* Both genders will be recruited; At least 10% of participants will be men. Enrollment of women will be capped at n = 324 (90%) to meet this goal.
* All ethnic groups will be recruited, with a goal of recruiting 10% minorities
* English speaking
* Have access to the Internet via a computer, and basic computer skills

Exclusion Criteria:

* Report health problems that make weight loss or unsupervised exercise unsafe or unreasonable
* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire1
* Are currently pregnant or breastfeeding, or intend to become pregnant in the next 12 months
* Are planning to move outside of the state within the next 12 months
* Report any cognitive or physical limitations that preclude use of a personal computer
* Have participated in a study conducted by the WCDRC or UT in the past 2 years
* Have followed a commercial weight-loss program within the previous 6 months or who are currently following a commercial weight loss program
* Weight loss of ≥ 5% of initial body weight in the last 6 months
* History of clinically diagnosed eating disorder excluding Binge Eating Disorder.
* Previous surgical procedure for weight loss
* Currently taking weight loss medication
* Treatment of cancer within the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in body weight, measured in kilograms | 3 and 6 months after randomization

SECONDARY OUTCOMES:
Engagement with the electronic intervention system, measured by number of body weights, foods, and physical activity bouts recorded per week | 3 and 6 months after randomization

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Weight Control and Diabetes Resarch Center, Providence, Rhode Island
  - University of Tennessee, Knoxville, Tennessee